CLINICAL TRIAL: NCT05068934
Title: The Relationship Between Epicardial Fat Tissue and Cardiac Function in HFpEF
Brief Title: The Relationship Between Epicardial Fat Tissue and Cardiac Function in HFpEF Patients
Status: Completed | Type: Observational
Sponsor: Dongying Zhang (Other)
Responsible Party: Sponsor-Investigator, Dongying Zhang, Dongying Zhang, Chongqing Medical University
Organization: Chongqing Medical University (Other)
Other Study IDs: 2020-09
Record Dates: First submitted 2021-09-26; First posted 2021-10-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: Epicardial Adipose tissue; Cardiac Function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Heart failure with preserved ejection fraction (HFpEF) refers to a group of symptoms and signs of heart failure, normal or near-normal left ventricular systolic function (EF>50%), and ventricular muscle diastolic dysfunction and A clinical syndrome characterized by decreased compliance and increased stiffness. The pathogenesis of HFpEF is related to impaired lipid metabolism and inflammation. Epicardial adipose tissue (Epicardial Adipose tissue, EAT) is a kind of visceral adipose tissue. Related studies have shown that extracardiac Membrane fat is related to inflammation markers, cardiometabolic risk and cardiovascular disease.However, there is still no research investigating the the relationship between epicardial fat thickness and Cardiac Function in HFpEF patients.

DETAILED DESCRIPTION:
Heart failure with preserved ejection fraction (HFpEF) refers to a group of symptoms and signs of heart failure, normal or near-normal left ventricular systolic function (EF>50%), and ventricular muscle diastolic dysfunction and A clinical syndrome characterized by decreased compliance and increased stiffness. The pathogenesis of HFpEF is related to impaired lipid metabolism and inflammation. Epicardial adipose tissue (Epicardial Adipose tissue, EAT) is a kind of visceral adipose tissue, which is composed of adipose tissue deposited between the myocardium and the visceral layer of the pericardium. It is closely adjacent to the coronary arteries and myocardium. Related studies have shown that extracardiac Membrane fat is related to inflammation markers, cardiometabolic risk and cardiovascular disease.However, there is still no research investigating the the relationship between epicardial fat thickness and Cardiac Function in HFpEF patients. This study intends to observe the relationship between epicardial fat thickness and left and right functions in patients with HFpEF, and evaluate whether epicardial fat thickness can be used as an indicator of left and right dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged >=18years old;
* Diagnosed with HFpEF.

Diagnostic criteria including:

1. left ventricular ejection fraction ≥50%；
2. with the symptoms and/or signs of heart failure；
3. BNP≥35 pg/mL and/or NTproBNP≥125 pg/mL；
4. at least one additional criterion: relevant structural heart disease(LVH and/or LAE) or diastolic dysfunction

Exclusion Criteria:

* LVEF less than 45% at any time;
* Severe liver failure;
* Primary pulmonary hypertension;
* Age <18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients with preserved ejection fraction (HFpEF)
Sampling Method: Non-Probability Sample
Enrollment: 1083 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Epicardial Fat Tissue | On admission
  Epicardial Fat Tissue by cardiac color Doppler ultrasound
Cardiac Function | On admission
  Left ventricular diastolic function and right ventricular systolic function by cardiac color Doppler ultrasound
Composite Endpoint of Worsening Heart Failure Event and Cardiovascular Death | From date of discharge until the date of first worsening HF event or date of death, whichever came first, assessed up to 5 years
  Composite Endpoint of Worsening Heart Failure Event and Cardiovascular Death

SECONDARY OUTCOMES:
Worsening HF Event | From date of discharge until the date of first worsening HF event or date of death, whichever came first, assessed up to 5 years
  Worsening Heart Failure Event
CV Death | From date of discharge until the date of death, whichever came first, assessed up to 10 years
  Cardiovascular Death
All-cause Death | From date of discharge until the date of death, whichever came first, assessed up to 10 years
  Death from any causes

CONTACTS AND LOCATIONS:
Overall Officials: Dongying Zhang, doctor, Study Director — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: No